CLINICAL TRIAL: NCT03943290
Title: An Open-Label Extension Study to Evaluate the Long-Term Effects of ACE-083 in Patients With Facioscapulohumeral Muscular Dystrophy (FSHD) Previously Enrolled in Study A083-02 and in Patients With Charcot-Marie Tooth (CMT) Disease Types 1 and X Previously Enrolled in Study A083-03
Brief Title: Extension Study to Evaluate the Long-Term Effects of ACE-083 in Patients With Facioscapulohumeral Muscular Dystrophy (FSHD) and Charcot-Marie Tooth (CMT) Disease Types 1 and X (CMT1 and CMTX)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigation of ACE-083 for use in patients with CMT and FSHD is being discontinued in this extension study as functional secondary endpoints were not achieved in the A083-023 or A083-03 trial (the parent trials).
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A083-04; ACE-083 (Other: Acceleron Pharma Inc.)
Record Dates: First submitted 2019-04-17; First posted 2019-05-09 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Facioscapulohumeral Muscular Dystrophy; Charcot-Marie-Tooth Disease
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1 Cohort 1a (Experimental): ACE-083 240 mg/muscle administered bilaterally by injection into the TA muscle every 4 weeks for up to 6 doses for FSHD patients
  Interventions: Drug: ACE-083
- Part 1 Cohort 1b (Experimental): ACE-083 240 mg/muscle administered bilaterally by injection into the BB muscle every 4 weeks for up to 6 doses for FSHD patients
  Interventions: Drug: ACE-083
- Part 1 Cohort 1c (Experimental): ACE-083 240 mg/muscle administered bilaterally by injection into the TA muscle every 4 weeks for up to 6 doses for CMT patients
  Interventions: Drug: ACE-083
- Part 2 Cohort 2a (Experimental): ACE-083 Administered into the TA muscle q4w for up to 24 months (24 doses) for FSHD patients
  Interventions: Drug: ACE-083
- Part 2 Cohort 2b (Experimental): ACE-083 Administered into the BB muscle q4w for up to 24 months (24 doses) for FSHD patients
  Interventions: Drug: ACE-083
- Part 2 Cohort 2c (Experimental): ACE-083 Administered into the TA muscle q4w for up to 24 months (24 doses) for CMT patients
  Interventions: Drug: ACE-083
- Part 2 Cohort 3a (Experimental): ACE-083 Administered into the TA muscle q8w for up to 24 months (12 doses) for FSHD patients
  Interventions: Drug: ACE-083
- Part 2 Cohort 3b (Experimental): ACE-083 Administered into the BB muscle q8w for up to 24 months (12 doses) for FSHD patients
  Interventions: Drug: ACE-083
- Part 2 Cohort 3c (Experimental): ACE-083 Administered into the TA muscle q8w for up to 24 months (12 doses) for CMT patients
  Interventions: Drug: ACE-083

INTERVENTIONS:
Drug: ACE-083 — Recombinant fusion protein

SUMMARY:
This is an open-label, multicenter, phase 2 extension study to evaluate the safety, tolerability, PK, PD, and efficacy of ACE-083 in subjects with FSHD previously enrolled in Study A083-02 and subjects with CMT1 and CMTX previously enrolled in Study A083-03. This study will be conducted in two Parts: Part 1, which is a loading phase of 6 months' duration, and Part 2, the maintenance phase, which will last up to 24 months.

DETAILED DESCRIPTION:
Part 1 (6-month, non-randomized, open-label, loading phase for subjects from A083-02 Part 1 and A083-03 Part 1) Part 1 will consist of 3 cohorts of up to 18 subjects each. Subjects enrolled in Cohorts 1a and 1b will have completed Part 1 of Study A083-02; subjects enrolled in Cohort 1c will have completed Part 1 of Study A083-03. In this loading phase, 240 mg/muscle ACE-083 will be administered bilaterally every 4 weeks (q4w) for 6 doses (6 months) into either the tibialis anterior (TA) muscle or the biceps brachii (BB) muscle, depending on the muscle injected in the previous study; subjects may not switch muscle cohort upon enrollment in this study. Subjects will participate in a screening period of up to 4 weeks before receiving the first dose of ACE-083.

Part 2 (24-month, randomized, open-label rollover maintenance phase for subjects from A083-02 Part 2, A083-03 Part 2, and A083-04 Part 1) Subjects who complete Part 1 of this study (the loading phase), Part 2 of A083-02, or Part 2 of A083-03 will enroll directly into the Part 2 open-label maintenance phase of treatment with ACE-083 and will consist of 6 cohorts of up to 23 FSHD or 29 CMT subjects each. These subjects will be randomized (1:1) to receive ACE-083, 240 mg/muscle bilaterally, either q4w or q8w. Thus, subjects enrolled in Cohorts 2a, 2b, and 2c will be FSHD TA, FSHD BB, and CMT TA treated q4w, and subjects enrolled in Cohorts 3a, 3b, and 3c will be FSHD TA, FSHD BB, and CMT TA treated q8w.

Study duration for a subject initially enrolled in Part 1 and then extended to Part 2 will be approximately 33 months, including a 1-month screening period, 6-month Part 1 loading phase, 24-month Part 2 maintenance phase, and 2-month follow-up period.

For subjects who enrolled directly into Part 2 of this study from Part 2 of Studies A083-02 and A083-03, the duration of the study will be approximately 26 months, including a 24-month maintenance phase and a 2-month follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Completion of treatment with study drug per protocol and completion of the end of treatment (ET) visit in Study A083-02 or Study A083-03.
2. Females of childbearing potential (defined as sexually mature women who have not undergone hysterectomy or bilateral oophorectomy or are not naturally postmenopausal ≥ 24 consecutive months) must have negative urine pregnancy test prior to enrollment and use highly effective birth control methods (abstinence, oral contraceptives, barrier method with spermicide, or surgical sterilization) during study participation and for 8 weeks following the last dose of ACE-083. Hormonal birth control use must be stable for at least 14 days prior to Day 1. Males must agree to use a condom during any sexual contact with females of childbearing potential while participating in the study and for 8 weeks following the last dose of ACE-083, even if they have undergone a vasectomy. Subjects must be counseled about contraception prior to the first dose of ACE-083 and every three months thereafter during the study.
3. Ability to adhere to the study visit schedule/procedures and to understand and comply with protocol requirements
4. Signed written informed consent

Key Exclusion Criteria:

1. Current/active malignancy (e.g., remission less than 5 years' duration), with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
2. Co-morbidities, including symptomatic cardiopulmonary disease, significant orthopedic or neuropathic pain, or other conditions that, in the opinion of the investigator, would limit a subject's ability to complete strength and/or functional assessments
3. Type 1 or type 2 diabetes mellitus
4. Thyroid disorder unless condition is stable with no change in treatment for at least 4 weeks before the first dose and no expected change for duration of study
5. Renal impairment (serum creatinine ≥ 2 times the upper limit of normal [ULN])
6. Aspartate transaminase (AST) and/or alanine transaminase (ALT) ≥ 3 times ULN
7. Increased risk of bleeding (i.e., due to hemophilia, platelet disorders, or use of any anticoagulation/platelet modifying therapies up to 2 weeks prior to Study Day 1 and for duration of study; single agent low dose aspirin [≤ 100 mg daily] is permitted)
8. Severe deformity or ankle fixation that would sufficiently limit passive range of motion to affect functional assessments (TA patients only)
9. Major surgery within 4 weeks prior to Study Day 1
10. Chronic pharmacologic doses of systemic corticosteroids (≥ 2 weeks) within 4 weeks before Study Day 1 and for duration of study; intra-articular/topical/inhaled/intranasal physiologic doses of systemic corticosteroids are permitted
11. Androgens, growth hormone, insulin or oral hormone replacement therapy within 6 months before Study Day 1 and for duration of study; topical physiologic androgen replacement is permitted. Chronic insulin therapy is permitted for diabetic FSHD patients. Oral HRT is permitted if started at least 3 months prior to receiving study drug
12. Any change in medications potentially affecting muscle strength or function within 4 weeks of Study Day 1 and for duration of study (e.g., creatinine, CoQ10, systemic beta-adrenergic agonists)
13. Previous exposure to any other investigational agent (not including ACE-083) potentially affecting muscle volume, muscle strength, or muscle or nerve function within 5 half-lives of last dose plus an additional 8-week washout period (or 12 weeks prior to Study Day 1 if half-life is unknown)
14. Significant change in physical activity or exercise (e.g., significant increase or decrease in intensity or frequency) within 8 weeks before Study Day 1 or inability to maintain the baseline level of physical activity throughout the study
15. Any condition that would prevent MRI scanning or compromise the ability to obtain a clear and interpretable scan of the treated muscles (e.g., knee/hip replacement metallic implants)
16. Known active substance abuse, including alcohol
17. History of sensitivity to protein pharmaceuticals
18. Female that is pregnant or lactating/breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (19):
  - University of California-Irvine, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - Carolinas Healthcare System Neurosciences Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Montreal Neurological Institute & Hospital, Montreal, Quebec
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 Cohort 1a | Part 1 Cohort 1b | Part 1 Cohort 1c | Part 2 Cohort 2a | Part 2 Cohort 2b | Part 2 Cohort 2c | Part 2 Cohort 3a | Part 2 Cohort 3b | Part 2 Cohort 3c
Started | 7 | 1 | 13 | 6 | 7 | 6 | 6 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 1 | 13 | 6 | 7 | 6 | 6 | 8 | 8
Not completed — Sponsor Terminated Study | 6 | 1 | 11 | 6 | 7 | 6 | 6 | 7 | 8
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was used for baseline analysis- The Safety Population consisted of all participants enrolled/randomized in the study who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1a | Part 1 Cohort 1b | Part 1 Cohort 1c | Part 2 Cohort 2a | Part 2 Cohort 2b | Part 2 Cohort 2c | Part 2 Cohort 3a | Part 2 Cohort 3b | Part 2 Cohort 3c | Total
Number analyzed (Participants) | 7 | 1 | 13 | 6 | 7 | 6 | 6 | 8 | 8 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 13 | 5 | 6 | 5 | 6 | 8 | 8 | 59
  >=65 years | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (13.3) | 56 | 45.2 (15.5) | 51.7 (14.8) | 49.7 (14.6) | 55 (9.3) | 40.2 (14.3) | 40.4 (11.2) | 45.4 (10.7) | 46.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 7 | 4 | 2 | 3 | 5 | 2 | 5 | 32
  Male | 4 | 0 | 6 | 2 | 5 | 3 | 1 | 6 | 3 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 6 | 1 | 13 | 6 | 7 | 5 | 6 | 7 | 7 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 7 | 1 | 13 | 5 | 6 | 6 | 6 | 7 | 8 | 59
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 1 | 0 | 1 | 4 | 0 | 1 | 4 | 0 | 13
  United States | 5 | 0 | 13 | 3 | 2 | 6 | 3 | 2 | 8 | 42
  Spain | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Part 2- Frequency of Adverse Events - Presence and Nature of Adverse Events (AE) During Part 2
Description: The number of participants that had a least one Treatment Emergent Adverse Event during the Part 2 of the study. The pre-specified analysis for this outcome measure was for those participants in the part 2 cohorts of this study therefore, only data of part 2 portion of the study are reported.
Time Frame: From baseline to end of participation of the Part 2 portion of the study
Population: The Safety Population consisted of all participants enrolled/randomized in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2b | Part 2 Cohort 2c | Part 2 Cohort 3a | Part 2 Cohort 3b | Part 2 Cohort 3c
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8 | 8
Participants | 3 | 4 | 5 | 3 | 4 | 4

2. Primary Outcome: Part 2: Frequency of Adverse Events - Presence and Nature of Grade 3 or Higher Adverse Events (AE) During the Part 2 of the Study.
Description: The number of participants that had a least one grade 3 or higher Treatment Emergent Adverse Event during Part 2 of the study. The pre-specified analysis for this outcome measure was for those participants in the double-blind, placebo-controlled Part 2 of the study therefore, only data from the part 2 portion of the study are reported.
Time Frame: From baseline to the end of the part 2 portion of the study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2b | Part 2 Cohort 2c | Part 2 Cohort 3a | Part 2 Cohort 3b | Part 2 Cohort 3c
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 8 | 8
Participants | 0 | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Part 2: Change in Total Muscle Volume - Percent Change From Baseline to Day 113 in Total Muscle Volume of Injected Muscle by Magnetic Resonance Imaging (MRI) During the Part 2 Portion
Description: The primary pharmacodynamic variable was the difference in mean percent change in total muscle volume (average of left and right side) at the first 6 months of the maintenance phase (Day 169; q4w or q8w) from the total muscle volume (average of left and right sides) at the start of the maintenance phase (or equivalently the end of the loading phase). Due to the early termination of this trial, percent change is only able to be reported as percent change from baseline to Day 113. The pre-specified analysis for this outcome measure was for those participants in the part 2 portion in cohorts with data to Day 113. Therefore, only data from these part 2 arms- 2b, 2c, 3b and 3c of the study are reported.
Time Frame: During the Part 2 portion of the study: Baseline to Day 113
Population: Per Protocol Set (PPS) consisted of all participants enrolled/randomized in the study, who received at least 1 dose of study drug with no clinical study report-reportable protocol violations and at least 1 post-baseline MRI evaluation.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part 2 Cohort 2b | Part 2 Cohort 2c | Part 2 Cohort 3b | Part 2 Cohort 3c
Number analyzed (Participants) | 2 | 3 | 1 | 3
percent change | 6.49 (8.63) | 19.36 (13.78) | -12.14 | 12.72 (1.18)

4. Secondary Outcome: Part 2: Change in Muscle Function. Absolute Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle:10-meter Walk/Run During Part 2 of the Study
Description: Timing (in seconds) participants took to complete a 10-meter walk/run distance. Baseline and end of treatment visit values were used to report absolute change from baseline in functional assessment due to early termination of the trial. The pre-specified analysis for this outcome measure was for those participants with data available at baseline and at the end of treatment in part 2 of this study therefore, only data from the part 2 cohorts 2a, 2c and 3a of the study are reported.
Time Frame: Baseline and End of Treatment visit for Part 2 of the study
Population: Per Protocol Set: All patients enrolled/randomized in the study who have received at least one dose of study drug (includes placebo) with no major protocol violations.
Measure: Mean (Standard Error); unit: seconds
Groups:
- Part 2 Cohort 2a: ACE-083 Administered into the TA muscle q4w for up to 24 months (24 doses) for FSHD patients ACE-083: Recombinant fusion protein
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2c | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 1 | 6
seconds | 0.5 (0.38) | -0.4 | 0.3 (0.51)

5. Secondary Outcome: Part 2: Change in Muscle Function. Percent Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle:10-meter Walk/Run During Part 2 of the Study
Description: as for outcome 4
Time Frame: Baseline and End of Treatment visit for Part 2 of the study
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2c | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 1 | 6
percent change | 5.29 (4.05) | -5.06 | 2.55 (5.45)

6. Secondary Outcome: Part 2: Change in Muscle Function. Absolute Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle: 6-minute Walk Test
Description: During Part 2: for the 6-minute walk test, participants walked at normal pace for six minutes and the distance was measured in meters. Absolute change from baseline to end of treatment in phase 2 were reported since this trial was terminated early. Further, only part 2 cohorts 2a, 2c, and 3a had data to report for this analysis.
Time Frame: Baseline and End of Treatment Visit during Part 2 of the study
Population: as for outcome 3
Measure: Mean (Standard Error); unit: meters
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2c | Part 2 Cohort 3a
Number analyzed (Participants) | 4 | 1 | 5
meters | 12.25 (17.3) | 14 | 0 (7.44)

7. Secondary Outcome: Part 2: Change in Muscle Function - Percent Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle in 6-minute Walk Test
Description: During Part 2: for the 6-minute walk test, participants walked at normal pace for six minutes and the distance was measured in meters. Absolute change from baseline to end of treatment in phase 2 were reported since this trial was terminated early. Further, only part 2 cohorts 2a, 2c, and 3c had data to report for this analysis.
Time Frame: Baseline and End of Treatment visit during Part 2 of the study
Population: Per Protocol Set (PPS) consisted of all participants enrolled/randomized in the study, who received at least 1 dose of study drug with no clinical study report-reportable protocol violations.
Measure: Mean (Standard Error); unit: percent change
Groups:
- Part 2 Cohort 3c: ACE-083 Administered into the TA muscle q8w for up to 24 months (12 doses) for FSHD patients ACE-083: Recombinant fusion protein
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2c | Part 2 Cohort 3c
Number analyzed (Participants) | 4 | 1 | 5
percent change | 4.46 (4.27) | 3.82 | -0.39 (2.23)

8. Secondary Outcome: Part 2: Change in Muscle Function. Absolute Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle: 4-stair Climb Up (in Participants With FSHD Only)
Description: During Part 2 in FSHD participants only: This is a measure (in seconds) of participants going up 4 standard stairs. Absolute Change is compared from baseline to the end of treatment visit as this trial was terminated early. As this analysis was pre-specified for FSHD patients only, data is only reported for participants with FSHD (cohorts 2a and 3a).
Time Frame: Baseline, End of Treatment visit during Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 6
seconds | -0.16 (0.38) | -0.5 (0.34)

9. Secondary Outcome: Part 2: Change in Muscle Function - Percent Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle in 4-stair Climb Up (in Participants With FSHD Only)
Description: During Part 2 in FSHD participants only: This is a measure (in seconds) of participants going up 4 standard stairs. Percent Change is compared from baseline to the end of treatment visit as this trial was terminated early. As this analysis was pre-specified for FSHD patients only, data is only reported for participants with FSHD (cohorts 2a and 3a).
Time Frame: Baseline, End of Treatment visit during Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 6
percent change | 2.78 (9.10) | -7.58 (4.51)

10. Secondary Outcome: Part 2: Change in Muscle Function. Absolute Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle: 4-stair Climb Down (in Participants With FSHD Only)
Description: During Part 2 (in FSHD participants only)This is a measure (in seconds) of participants going down 4 standard stairs. Absolute Change is compared from baseline to the end of treatment visit as this trial was terminated early. As this analysis was pre-specified for FSHD patients only, data is only reported for participants with FSHD (cohorts 2a and 3a).
Time Frame: Baseline, End of Treatment visit during Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 6
seconds | 0.74 (0.77) | -0.18 (0.22)

11. Secondary Outcome: Part 2: Change in Muscle Function. Percent Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle: 4-stair Climb Down (in Patients With FSHD Only)
Description: During Part 2 (in FSHD participants only)This is a measure (in seconds) of participants going down 4 standard stairs. Percent Change is compared from baseline to the end of treatment visit as this trial was terminated early. As this analysis was pre-specified for FSHD patients only, data is only reported for participants with FSHD (cohorts 2a and 3a).
Time Frame: Baseline, End of Treatment visit during Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 6
percent change | 6.81 (7.72) | -6.89 (5.19)

12. Secondary Outcome: Part 2: Change in Muscle Function. Absolute Change From Baseline in Functional Assessment for Tibialis Anterior (TA) Muscle: 100-meter Timed Test
Description: During Part 2 this measure is the timing (in seconds) to complete 100-meter walk test. Percent Change is reported from baseline to the end of treatment visit as this trial was terminated early. As this analysis was pre-specified for part 2 only, data is only reported for participants with FSHD and CMT in part 2 with data for both timepoints (cohorts 2a, 2c and 3a).
Time Frame: Baseline, End of Treatment visit for Part 2 of the study
Population: as for outcome 7
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2c | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 1 | 6
seconds | 6.8 (3.64) | 10 | 8.8 (5.78)

13. Secondary Outcome: Part 2: Change in Muscle Function - Percent Change From Baseline for Tibialis Anterior (TA) Muscle in 100-meter Timed Test
Description: as for outcome 12
Time Frame: Baseline, End of Treatment visit, Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2c | Part 2 Cohort 3a
Number analyzed (Participants) | 5 | 1 | 6
percent change | 8.49 (3.68) | 13.51 | 14.82 (12.41)

14. Secondary Outcome: Part 2: Change in Muscle Function. Absolute Change From Baseline in Functional Assessment for Biceps Brachii (BB) Muscle: Mid-level Performance of the Upper Limb (PUL) Test.
Description: Part 2: Performance of upper limb (PUL) - Middle level elbow dimension score- Sum of the 9 items for this particular dimension (Minimum=0, Maximum = 34, with higher scores indicating increased functionality). These include: "Hand(s) to Mouth", "Hand(s) to table from lap", "Move weight on table", "Lifting light cans", "Lifting heavy cans", "Stacking light cans", "Stacking heavy cans", "Remove lid from container", and "Tearing paper". Pre-specified analysis was for absolute change in BB cohorts for FSHD participants only with Baseline and End of Treatment visit data (cohorts 2b and 3b) due to the early termination of the study. Thus, data is only reported for these two cohorts.
Time Frame: Baseline, End of Treatment visit during Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2 Cohort 2b | Part 2 Cohort 3b
Number analyzed (Participants) | 6 | 7
units on a scale | 0.5 (0.34) | 0 (0)

15. Secondary Outcome: Part 2: Change in Muscle Function - Percent Change From Baseline for Biceps Brachii (BB) Muscle in Mid-level Performance of the Upper Limb (PUL) Test
Description: Part 2: Performance of upper limb (PUL) - Middle level elbow dimension score- Sum of the 9 items for this particular dimension (Minimum=0, Maximum = 34, with higher scores indicating increased functionality). These include: "Hand(s) to Mouth", "Hand(s) to table from lap", "Move weight on table", "Lifting light cans", "Lifting heavy cans", "Stacking light cans", "Stacking heavy cans", "Remove lid from container", and "Tearing paper". Pre-specified analysis was for percent change in BB cohorts for FSHD participants only with Baseline and End of Treatment visit data (cohorts 2b and 3b) due to the early termination of the study. Thus, data is only reported for these two cohorts.
Time Frame: Baseline, End of Treatment
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percent change in units on scale
Arm/Group | Part 2 Cohort 2b | Part 2 Cohort 3b
Number analyzed (Participants) | 6 | 7
percent change in units on scale | 1.55 (1.06) | 0 (0)

16. Secondary Outcome: Part 2: Change in Muscle Function. Absolute Change From Baseline in Functional Assessment for Biceps Brachii (BB) Muscle: Upper Level Performance of the Upper Limb (PUL) Test.
Description: Performance of upper limb (PUL) -PUL upper level/shoulder dimension- Shoulder domain score which represents the sum of the following 4 items that the patient is asked to do on the preferred side [either right or left side identified by patient to be done on the same side for all scheduled times]: a. Largest weight patient can use to perform shoulder abduction to shoulder height (elbow to shoulder level) b. Largest weight patient can use to perform shoulder abduction above shoulder height (elbow to eye level) c. Largest weight patient can use to perform shoulder flexion to shoulder height (elbow to shoulder level) d. Largest weight patient can use to perform shoulder flexion above shoulder height (elbow to eye level) Each of the 4 components above is scored depending on the highest weight performed where scores are: 0 = Unable; 1 = Able no weights; 2 = 200 g; 3 = 500 g; 4 = 1000 g. The maximum score is 16, with 16 being highest functionality. Reportable data is for Cohort 3b only.
Time Frame: Baseline, End of Treatment visit during part 2 of the study
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2 Cohort 3b
Number analyzed (Participants) | 4
units on a scale | 3.75 (3.75)

17. Secondary Outcome: Part 2: Change in Muscle Function. Percent Change From Baseline in Functional Assessment for Biceps Brachii (BB) Muscle: Upper Level Performance of the Upper Limb (PUL) Test.
Description: as for outcome 16
Time Frame: Baseline, End of Treatment visit during Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: percent change units on a scale
Arm/Group | Part 2 Cohort 3b
Number analyzed (Participants) | 4
percent change units on a scale | 375 (375)

18. Secondary Outcome: Part 2: Change in Patient-reported Quality of Life. Absolute Change From Baseline in FSHD-health Index Total Score (FSHD-HI, in Patients With FSHD Only)
Description: The FSHD Health Index (FSHD-HI) is a disease-specific patient reported outcome questionnaire that uses direct patient input to measure disease burden. For this index, the total score is scored from 0 to 100 with 0 representing no disease burden and 100 representing the maximum amount of disease burden in the particular domain. Pre-specified analysis was for FSHD cohorts only with absolute change in total score reported as this trial was terminated early.
Time Frame: Baseline, End of Treatment visit during part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2 Cohort 2a | Part 2 Cohort 2b | Part 2 Cohort 3a | Part 2 Cohort 3b
Number analyzed (Participants) | 1 | 6 | 4 | 3
units on a scale | -0.39 | -1.14 (2.53) | -2.63 (1.74) | 0.80 (4.19)

19. Secondary Outcome: Part2: Change in Patient-reported Quality of Life. Absolute Change From Baseline in CMT Health Index Total Score (CMT-HI, in Patients With CMT Only)
Description: Part 2: The CMT-Health Index (CMT-HI) is a disease-specific patient reported outcome measure designed to measure patient reported disease burden during clinical trials in patients with Charcot-Marie-Tooth Disease. For this index, the total score is scored from 0 to 100 with 0 representing no disease burden and 100 representing the maximum amount of disease burden. Pre-specified analysis was for cohorts of CMT participants only and due to the early termination of this trial, the absolute change is reported for the change from Baseline to Day 113.
Time Frame: Baseline, Day 113 during Part 2
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2 Cohort 2c | Part 2 Cohort 3c
Number analyzed (Participants) | 3 | 2
units on a scale | 9.72 (7.60) | -14.55 (9.99)

20. Secondary Outcome: Part 1: ACE-083 Serum Concentration Samples Part 1-Day1, 24-hour Post-dose
Description: Part1: ACE-083 serum concentration samples were taken on day 1, 24-hours post-dose. PK parameters of ACE-083 were not determined due to limited quantifiable concentration data. Pre-specified analysis was for part 1 cohorts only, therefore, available data is only reported for part 1 cohorts (1a, 1b and 1c). Mean and standard deviation descriptive statistics are being reported for the Day 1, 24-hour post-dose timepoint only, due to early termination of this trial.
Time Frame: day 1, 24 -hours post-dose in Part 1
Population: The PK Population consisted of all participants who received at least 1 dose of study drug and had sufficient PK samples collected and assayed for PK analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 Cohort 1a | Part 1 Cohort 1b | Part 1 Cohort 1c
Number analyzed (Participants) | 7 | 1 | 13
ng/mL | 38.3 (13.8) | 76.4 | 41.10 (12.6)

21. Secondary Outcome: Part1: ACE-083 Serum Concentration Samples Part 1-Day 85, 24-hour Post-dose
Description: Part1: ACE-083 serum concentration samples were taken on day 85, 24-hours post-dose. PK parameters of ACE-083 were not determined due to limited quantifiable concentration data. Pre-specified analysis was for part 1 cohorts only, therefore, available data is only reported for part 1 cohorts (1a, 1b and 1c). Mean and standard deviation descriptive statistics are being reported for the Day 85, 24-hour post-dose timepoint only, due to early termination of this trial.
Time Frame: day 85, 24 -hours post-dose in Part 1
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 Cohort 1a | Part 1 Cohort 1b | Part 1 Cohort 1c
Number analyzed (Participants) | 7 | 1 | 13
ng/mL | 23.1 (2.26) | 53 | 39.34 (18.2)

22. Secondary Outcome: Part1: Pharmacokinetics Parameter of Time to Maximum Serum Concentration Following Administration (Tmax)
Description: Part 1: ACE-083 concentrations ranged from 20.1 to 238.6 μg/L across FSHD and CMT cohorts with the majority of serum concentrations were below the lower limit of quantification (LLOQ) or just above LLOQ. Further, given the early termination of this trial, there were not enough samples per cohort collected at the pre-specified timeline points to be able to determine Tmax.
Time Frame: From baseline to End of Treatment in Part 1
Population: as for outcome 20
Arm/Group | Part 1 Cohort 1a | Part 1 Cohort 1b | Part 1 Cohort 1c
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Part1: Pharmacokinetics Parameter of Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Part 1: ACE-083 concentrations ranged from 20.1 to 238.6 μg/L across FSHD and CMT cohorts with the majority of serum concentrations were below the lower limit of quantification (LLOQ) or just above LLOQ. Further, given the early termination of this trial, there were not enough samples per cohort collected at the pre-specified timeline points to be able to determine AUC.
Time Frame: From baseline to End of Treatment in Part 1
Population: as for outcome 20
Arm/Group | Part 1 Cohort 1a | Part 1 Cohort 1b | Part 1 Cohort 1c
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For Part 1, adverse event data was collected for six months from baseline. For Part 2, adverse event data was collected for 24 months from baseline.
Arm/Group | Part 1 Cohort 1a | Part 1 Cohort 1b | Part 1 Cohort 1c | Part 2 Cohort 2a | Part 2 Cohort 2b | Part 2 Cohort 2c | Part 2 Cohort 3a | Part 2 Cohort 3b | Part 2 Cohort 3c
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/1 | 0/13 | 0/6 | 0/7 | 0/6 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/1 | 0/13 | 0/6 | 0/7 | 0/6 | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/7 | 1/1 | 11/13 | 3/6 | 4/7 | 5/6 | 3/6 | 4/8 | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1a (N=7) | Part 1 Cohort 1b (N=1) | Part 1 Cohort 1c (N=13) | Part 2 Cohort 2a (N=6) | Part 2 Cohort 2b (N=7) | Part 2 Cohort 2c (N=6) | Part 2 Cohort 3a (N=6) | Part 2 Cohort 3b (N=8) | Part 2 Cohort 3c (N=8)
injection site bruising (General disorders) | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0
injection site discomfort (General disorders) | 0 | 0 | 6 | 0 | 0 | 1 | 0 | 1 | 0
injection site erythema (General disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 2 | 1
injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
injection site pain (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
injection site papule (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
injection site pruritus (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
injection site swelling (General disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1
injection site warmth (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
vessel puncture site bruise (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0
sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
hypersensivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
atrioventricular block first degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
c-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
In this open-label, multicenter, phase 2 extension study in participants with FSHD and CMT (types 1 and X), treatment with ACE-083 q4w or q8w was generally safe and well tolerated. Participants were discontinued from this study when their respective parent studies were terminated by the sponsor, and as such, this study was also terminated. Due to premature termination of this study, insufficient efficacy data were obtained to enable meaningful efficacy analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03943290/Prot_000.pdf